CLINICAL TRIAL: NCT01549236
Title: Population Pharmacokinetics Study of Benznidazole in Children With Chagas'Disease
Acronym: Pop PK Chagas
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Drugs for Neglected Diseases (Other)
Collaborators: LAT Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DNDi-CD-PEDBZ-001
Record Dates: First submitted 2012-03-01; First posted 2012-03-09 (Estimated); Last update posted 2018-06-25 (Actual); Status verified 2012-08

CONDITIONS: Chagas' Disease
Keywords: Chagas Disease; Trypanosoma Cruzi; T.Cruzi
MeSH Terms: conditions — Chagas Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Benznidazole 12,5mg or 100mg — All 80 subjects recruited into the study will receive treatment with:
  - Benznidazole (Laboratório Farmacêutico do Estado de Pernambuco -LAFEPE - Recife - Brazil; tablet 12.5mg or 100mg), 7.5 mg/Kg/day PO (actual range of 5.5-8.5 mg/Kg/d), divided in two daily doses, for 60 days.
  Other Names: BNZ

SUMMARY:
The purpose of this study is to describe the population pharmacokinetics parameters of benznidazole in children with acute or early chronic indeterminate form of Chagas Disease.

DETAILED DESCRIPTION:
Treatment of Chagas disease (CD) has been always focused on pediatric population. Initially, treatment was recommended only to acute and congenital cases (including newborns diagnosed at birth), with good parasitological response of 60% to 85% of patients in the acute phase and more than 90% of congenitally infected infants treated in the first year of life.

Despite existing treatment recommendations for children with CD (from birth to 12y), there is no formulation available that meets the needs of target pediatric population, especially the younger age groups. Benznidazole (Bz), developed over 30 years ago and the main drug of choice, is only available in an 'adult' tablet strength of 100 mg (LAFEPE Benznidazol®).

With the lack of pediatric formulation, the 100mg tablet needs to be fractionated in ½ and ¼ tablets or prepared as extemporaneous formulations (macerated, diluted, suspension, etc) to adjust the dose to patient weight, often leading to sub or over-dosing, which may affect safety and efficacy of the treatment. With regards to children, there is an absolute lack of information on Bz PK in the pediatric population and its relationship with treatment safety and efficacy.

In order to respond to the need of a age-adapted, easy to use pediatric formulation, DNDi and LAFEPE have joined efforts to develop a 12.5 mg dispersible Bz tablet targeting treatment of CD in children < 20 Kg. Once this formulation is available, two pharmacokinetics studies are planned to be conducted: a comparative bioavailability study in adult healthy normal volunteers and a population pharmacokinetics study in young children.

The group of newborns, from birth to - 2 years-old children, has been included as they represent the population of congenital cases. Current estimates of positive serology for CD in women at reproductive age vary considerably from country-to-country ranging from 5-40%, with vertical transmission rates of up to 12%. There is consensus that congenital infection may remain an important mode of transmission for another generation, and appropriate treatment targeting newborns is a possible control strategy (with very high chances of cure) with the new pediatric formulation.

Children 2-12 years-old have also been included as a target population, to represent those who may have been infected via congenital or vector-borne transmission, and usually present with the early chronic indeterminate form of the disease. In CD endemic countries these groups of children are usually diagnosed through school or community screening programs, and also have a high chance of cure (> 60-75%) with Bz treatment.

Population PK has been chosen as the study design as it would minimise the number of samples per patient, an important requirement for studies conducted in the pediatric population. The dearth of PK data in adults and lack of information on the variability in the target population does not allow for power calculations and the use of optimal sampling design for definition of the timing of samples. Experts reviewed the available information and recommended sparse sampling, with 5 PK samples distributed over the absorption phase (1 sample), steady-state (2 samples) and elimination phase (2 samples). With a total of 5 PK measurements per patient and a total of 80 patients stratified by age, it is expected that PK curves and variability can be drawn with an adequate level of precision.

PK data obtained from this study is expected to inform an age-adapted Bz regimen for the pediatric population affected by CD.

ELIGIBILITY:
Inclusion Criteria:

* Age between newborn (1day) - 12 years
* Diagnosis of T. cruzi infection by:

  * Direct microscopic examination or
  * Conventional serology, at least two positive tests (ELISA, IIF or HAI)
* Written informed consent form by parent/ legal representative
* Children assent if > 7 years

Exclusion Criteria:

* Pre-term (< 37 weeks gestational age) or weight < 2500 g
* Female subject who has reached menarche
* Subjects presenting any other acute or chronic health conditions, that in the opinion of the PI, may interfere with the PK, efficacy and/or safety evaluation of the study drug
* Known history of hypersensitivity or serious adverse reactions to nitro- imidazoles
* History of CD treatment with benznidazole or nifurtimox in the past
* Immunocompromised patients (clinical history compatible with HIV infection, primary immunodeficiency or prolonged treatment with corticosteroids or other immunosuppressive drugs)
* Abnormal laboratory test values at screening for the following parameters: total WBC count, platelet count, ALT, AST, total bilirubin and creatinine.

Exception for this criterion is considered for newborns with congenital Chagas Disease, for whom ALT/AST and bilirubin will not be considered exclusion criteria unless considered clinically significant by the investigator.

* Inability to comply with follow-up and/or not having a permanent address
* Any condition that prevents the subject from taking oral medication

Ages: 1 Day to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2011-05 (Actual); Primary Completion 2012-08 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics Endpoints | Day 60
  Plasma level concentrations of benznidazol determined in children at first day of treatment (Day 0), steady state phase (D7 and Day 30) and at the end of treatment (Day 60).
  Population pharmacokinetics parameters of benznidazole in children, including CL, Vd, and Ka.
  Individual AUC.
  Individual Cmax.
  Individual Cmin.
  Individual t1/2 will be estimated using population parameters.

SECONDARY OUTCOMES:
Efficacy Endpoints | Day 60
  Parasitological cure rate as determined by qualitative PCR at the end of treatment (Day 60).
Safety endpoints | Day 60
  Rate of Serious of Adverse Events and/or adverse events leading to treatment discontinuation.
Safety Endpoints | Day 60
  Rate and severity of adverse events.
  Covariates to be evaluated: age, gender, weight, height, parasite load at baseline and phase of disease (acute vs chronic).

CONTACTS AND LOCATIONS:
Overall Officials: Jaime Altcheh, MD, Principal Investigator — Argentina: FIPEC Foundation (Fundación para el Estudio de las Infecciones Parasitarias y Enfermedad de Chagas
Locations (3):
- Argentina (3):
  - Hospital General de Niños Ricardo Gutierrez, Buenos Aires
  - Hospital Público Materno Infantil, Salta
  - Hospital de Niños "Doctor Héctor Quintana", San Salvador de Jujuy

REFERENCES:
- [Background] Andrade AL, Martelli CM, Oliveira RM, Silva SA, Aires AI, Soussumi LM, Covas DT, Silva LS, Andrade JG, Travassos LR, Almeida IC. Short report: benznidazole efficacy among Trypanosoma cruzi-infected adolescents after a six-year follow-up. Am J Trop Med Hyg. 2004 Nov;71(5):594-7. PMID 15569790
- [Background] de Andrade AL, Zicker F, de Oliveira RM, Almeida Silva S, Luquetti A, Travassos LR, Almeida IC, de Andrade SS, de Andrade JG, Martelli CM. Randomised trial of efficacy of benznidazole in treatment of early Trypanosoma cruzi infection. Lancet. 1996 Nov 23;348(9039):1407-13. doi: 10.1016/s0140-6736(96)04128-1. PMID 8937280
- [Background] Sosa-Estani S, Segura EL. Etiological treatment in patients infected by Trypanosoma cruzi: experiences in Argentina. Curr Opin Infect Dis. 2006 Dec;19(6):583-7. doi: 10.1097/01.qco.0000247592.21295.a5. PMID 17075335
- [Background] Ribeiro I, Sevcsik AM, Alves F, Diap G, Don R, Harhay MO, Chang S, Pecoul B. New, improved treatments for Chagas disease: from the R&D pipeline to the patients. PLoS Negl Trop Dis. 2009 Jul 7;3(7):e484. doi: 10.1371/journal.pntd.0000484. No abstract available. PMID 19582163
- [Background] Garcia-Bournissen F, Altcheh J, Giglio N, Mastrantonio G, Della Vedova CO, Koren G. Pediatric clinical pharmacology studies in Chagas disease: focus on Argentina. Paediatr Drugs. 2009;11(1):33-7. doi: 10.2165/0148581-200911010-00012. PMID 19127950
- [Derived] Altcheh J, Moscatelli G, Caruso M, Moroni S, Bisio M, Miranda MR, Monla C, Vaina M, Valdez M, Moran L, Ramirez T, Patino OL, Riarte A, Gonzalez N, Fernandes J, Alves F, Ribeiro I, Garcia-Bournissen F. Population pharmacokinetics of benznidazole in neonates, infants and children using a new pediatric formulation. PLoS Negl Trop Dis. 2023 May 31;17(5):e0010850. doi: 10.1371/journal.pntd.0010850. eCollection 2023 May. PMID 37256863
- See also: Drugs for Neglected Diseases initiative — http://dndi.org